CLINICAL TRIAL: NCT01667757
Title: Angiographic and IVUS Criteria Defining Physiologic Optimization By the Fractional Flow Reserve After DES Implantation
Brief Title: Optimal Physiologic Intravascular Ultrasound Imaging Criteria After Drug Eluting Stent Implantation
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Joon Hyung Doh, MD, PHD, Inje University
Other Study IDs: IB-2-1208-026
Record Dates: First submitted 2012-08-12; First posted 2012-08-17 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Disease
Keywords: coronary atherosclerosis; drug eluting stent; intravascular ultrasound; fractional flow reserve
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- low post DES FFR group (<0.9): the patient with FFR values less than 0.9 after DES procedure
- high post DES FFR group (≥0.9): the patient with FFR values greater than 0.9 after DES procedure

SUMMARY:
Invasive imaging criteria of the Coronary arteriography (CAG) and intravascular ultrasound imaging (IVUS), satisfying procedural optimization after drug eluting stent (DES) implantation, were used in < 10% DS by CAG and 5-5.5mm2 MSA by IVUS. Whether these criteria satisfy not only relieving visible stenosis but also relieving lesion specific ischemia or not were unclear. Fractional flow reserve (FFR), an index of lesion specific ischemia, was proposed 0.9 as a physiologic criteria satisfying successful stent implantation by previous studies with bare metal stent. FFR after drug-eluting stent implantation can be an useful predictor for clinical outcome. But, direct comparative evaluation of the invasive imaging criteria defining as an indicator relieving myocardial ischemia were not reported. The aim of this study was to investigate angiographic and IVUS parameters in which corresponding FFR and evaluate their optimal physiologic criteria after DES implantation.

ELIGIBILITY:
Inclusion Criteria:

* clinical angina pectoris who underwent IVUS and FFR during coronary angiography and after DES implantation.
* agree with informed consent
* At least one segment of three major epicardial coronary arteries were consecutively enrolled in invasive CAG.
* Post- stent FFR and IVUS measurement performed at the immediately after whole PCI procedures.

Exclusion Criteria:

* unable to get informed consent
* low left ventricular ejection fraction less than 35%
* chronic renal failure (Cr > 2.0mg/dl)
* acute myocardial infarction related coronary artery
* allergy to adenosine injection

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent coronary angiography and percutaneous coronary intervention for the diagnosis and treatment purposes because of clinical angina pectoris. Patient who underwent simultaneous IVUS and FFR measurement after DES implantation would be enrolled consecutively.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Differences angiographic and IVUS parameters after DES between different FFR groups | baseline
  Angiographic residual percent diameter stenosis (%), minimal stent lumen diameter (mm) and total stent length (mm), and IVUS minimal stent cross-sectional area (mm2) and minimal stent lumen diameter (mm) will be compared according to different FFR groups at the time of measurement after DES implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Joon Hyung Doh, MDPhD, Principal Investigator — Inje University Ilsan Paik Hospital
Locations (1):
- Inje University Ilsan Paik Hospital, Goyang, Gyeonggido, South Korea

REFERENCES:
- [Background] Sonoda S, Morino Y, Ako J, Terashima M, Hassan AH, Bonneau HN, Leon MB, Moses JW, Yock PG, Honda Y, Kuntz RE, Fitzgerald PJ; SIRIUS Investigators. Impact of final stent dimensions on long-term results following sirolimus-eluting stent implantation: serial intravascular ultrasound analysis from the sirius trial. J Am Coll Cardiol. 2004 Jun 2;43(11):1959-63. doi: 10.1016/j.jacc.2004.01.044. PMID 15172398
- [Background] Doi H, Maehara A, Mintz GS, Yu A, Wang H, Mandinov L, Popma JJ, Ellis SG, Grube E, Dawkins KD, Weissman NJ, Turco MA, Ormiston JA, Stone GW. Impact of post-intervention minimal stent area on 9-month follow-up patency of paclitaxel-eluting stents: an integrated intravascular ultrasound analysis from the TAXUS IV, V, and VI and TAXUS ATLAS Workhorse, Long Lesion, and Direct Stent Trials. JACC Cardiovasc Interv. 2009 Dec;2(12):1269-75. doi: 10.1016/j.jcin.2009.10.005. PMID 20129555
- [Background] Nam CW, Rha SW, Koo BK, Doh JH, Chung WY, Yoon MH, Tahk SJ, Lee BK, Lee JB, Yoo KD, Cho YK, Chung IS, Hur SH, Kim KB, Choi CU, Oh DJ. Usefulness of coronary pressure measurement for functional evaluation of drug-eluting stent restenosis. Am J Cardiol. 2011 Jun 15;107(12):1783-6. doi: 10.1016/j.amjcard.2011.02.328. Epub 2011 Apr 8. PMID 21481824
- [Background] Nam CW, Hur SH, Cho YK, Park HS, Yoon HJ, Kim H, Chung IS, Kim YN, Kim KB, Doh JH, Koo BK, Tahk SJ, Fearon WF. Relation of fractional flow reserve after drug-eluting stent implantation to one-year outcomes. Am J Cardiol. 2011 Jun 15;107(12):1763-7. doi: 10.1016/j.amjcard.2011.02.329. Epub 2011 Apr 8. PMID 21481828